CLINICAL TRIAL: NCT04995185
Title: 18F-FMISO PET Guided Dose Escalation in Nasopharyngeal Carcinoma - a Feasibility and Planning Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Terry Fox Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MISSION16
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Hypoxia; FMISO; PET; Nasopharyngeal cancer
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Hypoxia; Nasopharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/CT imaging (Experimental): Intravenous injection of 370MBq ± 10% (18)F-fluoromisonidazole
  Interventions: Radiation: (18)F-fluoromisonidazole (FMISO)

INTERVENTIONS:
Radiation: (18)F-fluoromisonidazole (FMISO) — Patients do not need to be fasted prior to intravenous injection of 370MBq ± 10% (18)F-fluoromisonidazole. Scanning will be performed two hours after the injection. Patients will be scanned with their thermoplastic shell used in routine radiotherapy treatment for 10 minutes, followed by approximately 5 minutes scan of the upper chest.

SUMMARY:
This study aims to investigate the use of 18F-FMISO PET in identifying hypoxic subvolume for dose escalation radiotherapy in nasopharyngeal cancer and thus improve local control without significant increase in toxicities.

DETAILED DESCRIPTION:
The specific aims of this study are:

1. To establish hypoxia imaging in NPC patients
2. Investigate the dynamics of tumor hypoxia before and during chemoradiation
3. Integrate hypoxia imaging into radiation treatment planning protocols
4. Design hypoxia adapted radiation schedules
5. Identify candidate hypoxia biomarkers

ELIGIBILITY:
Inclusion Criteria:

* T3-T4 disease with no evidence of distant metastasis.
* Histological diagnosis of WHO Type II or III NPC
* No evidence of distant metastases in staging work up (including lung, liver and bone imaging).
* Planned for upfront radiotherapy and/or chemotherapy.
* Cross sectional imaging of the primary and neck disease (MRI preferred)
* Performance status of ECOG grade 0 or 1
* No prior tumour therapy
* At least 21 years of age, of either sex.
* Negative serum pregnancy test within 14 days prior to registration for women of childbearing potential;
* Adequate bone marrow, renal and hepatic function defined as follows:

Bone marrow: WBC > 3000 / mm3 (ANC > 1500 / mm3 ) Platelets > 100 000 / mm3. Hb > 10 gm/dl Renal: serum creatinine within institutional normal range(or) lower than the lower limit of institutional normal range : calculated creatinine clearance > 50 ml / min Hepatic: enzymes (SAP, SGOT) < 2x normal: bilirubin < 24 mol / l.

Exclusion Criteria:

* Allergic to 18F-fluoromisonidazole or Nitroimidazoles
* Planned for neoadjuvant chemotherapy
* Uncontrolled hypercalcaemia: calcium 2.7 mmol/L (10.8 mg/dL).
* Other serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator).
* Have serious active infection.
* Pregnant or lactating female subjects and subjects with reproductive potential not implementing adequate contraceptive measures

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
To investigate the dynamics of tumour hypoxia | From baseline and during 7 week long treatment regimen
  A repeat 18F-FMISO-PET in week 3 of the 7 weeks long treatment regimen is planned. Fractionated radiotherapy is expected to induce reoxygenation within the tumor as iterative process by killing well oxygenated tumor cells with every fraction thereby reducing oxygen demand in the remaining tumor cells. Repetitive hypoxia imaging at week 3 allows for assessment of evolution of hypoxia during radiotherapy.
To evaluate proportion of patients with contour-able hypoxic volume as well as the feasibility of generating dose-escalation radiotherapy plan with dosimetrically achieved parameters for target volume and organs-at-risk. | At baseline and week 3 of RT
  Number of patients with feasible radiotherapy plan dose-escalation to more than 84Gy
To estimate the correlation between immunohistochemical expression of CA-IX, VEGF and HIF-1a, (marker of hypoxia) and pre-treatment PET-SUV measurement | At baseline
To correlate 18F-FMISO PET uptake with tumor response at 3 months post radiotherapy, local control rate and disease free survival. | From baseline up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kiattisa Sommat, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - National Cancer Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No